CLINICAL TRIAL: NCT02327182
Title: A Long-Term Safety Study of MT-4666 in Patients With Mild to Moderate Alzheimer's Disease (AD)
Brief Title: Safety Study of MT-4666 in Subjects With Alzheimer's Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was terminated due to the benefit-risk balance of MT-4666.
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P211-05
Record Dates: First submitted 2014-12-23; First posted 2014-12-30 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Alzheimer's Disease
Keywords: MT-4666; α7 nicotinic acetylcholine receptor agonist; Alzheimer's Disease; Cognitive function; Dementia; Central Nervous System Agents
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MT-4666 low dose (Experimental): Low Dose, Tablet, Once Daily, For 52 Weeks
  Interventions: Drug: MT-4666
- MT-4666 high dose (Experimental): High Dose, Tablet, Once Daily, For 52 Weeks
  Interventions: Drug: MT-4666

INTERVENTIONS:
Drug: MT-4666

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of 2 fixed dose of MT-4666 administered once daily for 52 weeks with or without receiving a concomitant acetylcholinesterase inhibitors (AChEIs), in patients with mild to moderate Alzheimer's Disease (AD).

ELIGIBILITY:
Inclusion Criteria:

* Probable Alzheimer's disease consistent with the National Institute on Aging and the Alzheimer's Association Criteria for Diagnosis of Alzheimer's Disease (McKhann et al. 2011).
* MMSE score of ≥ 14 and ≤ 24 at the screening and ≥ 12 and ≤ 26 at the baseline.
* Modified Hachinski Ischemic Score (mHIS) ≤ 4 at the screening
* Appropriate caregiver available
* Subject living at home or in facilities who do not require continuous (24-hour) nursing care.

Exclusion Criteria:

* Diagnosis of any other disease which may cause dementia
* Diagnosis of major depressive disorder as defined by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) within last five years
* History of or current diagnosis of any psychosis
* History of myocardial infarction or unstable angina within six months before screening
* History of cerebrovascular disorder within 18 months before screening
* complication of hepatic disorder or renal dysfunction

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2014-12; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Safety of 2 fixed doses of EVP-6124 in subjects with Alzheimer's disease. Criteria for evaluation include: adverse events, clinical laboratory tests, vital signs, body weight, 12-lead ECG, Columbia Suicide Severity Rating Scale (C-SSRS) | Up to week 56

SECONDARY OUTCOMES:
Change in Mini Mental State Examination (MMSE) | baseline to Week 52
Change in Neuropsychiatric Inventory (NPI) total score | baseline to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Yu Nakamura, M.D., Ph.D., Study Director — Kagawa University School of Medicine; Kazuoki Kondo, M.D., Study Director — Tanabe Pharma Corporation
Locations (1):
- Investigational site, Osaka, Kansai, Japan